CLINICAL TRIAL: NCT01715467
Title: Community Registry Study Evaluating Dupuytren's Contracture Treatment. A Prospective, Observational, Longitudinal, Multicenter Study of the Treatment Patterns and Outcomes in Patients With Dupuytren's Contracture.
Brief Title: CORRECT: COmmunity RegistRy Study Evaluating Dupuytren's Contracture Treatment
Acronym: CORRECT
Status: Completed | Type: Observational
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: AUX-CC-901
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Dupuytren's Contracture
Keywords: Dupuytren; Contracture; Auxilium; XIAFLEX
MeSH Terms: conditions — Dupuytren Contracture; Contracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study will prospectively collect data on treatment options, patient/investigator satisfaction, requirement for retreatment or additional treatment, and long-term outcomes of 3 treatment modalities(XIAFLEX, fasciectomy, or fasciotomy/needle aponeurotomy) in patients with Dupuytren's contracture. In addition, this study will provide additional health economics and utilization data.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational study. Patients will be recruited based on the usual care presentation at each investigative site, as regular practice would dictate. Consecutive patients deemed eligible for the study by their physician will be invited to participate during their usual care visit. Enrolled patients will receive evaluations and treatment for Dupuytren's contracture according to the standard of care and clinical practice at each study site. No study-specific visits will be required as part of the study. Treatment and Follow-up Visits will be determined by the treating physician. Treatments received for Dupuytren's contracture will be recorded (ie, XIAFLEX, fasciectomy, or fasciotomy/needle aponeurotomy), including initial treatment and any subsequent therapy. The full prescribing information and medication guide for XIAFLEX is provided in this protocol as reference (Appendix B). Patient data (including treatment outcomes, joint contracture measured by the treating physician, and evidence of recurrence) and health care resource utilization data will be drawn from the patients' medical records, examination, and patient interviews. These data will be recorded via a web-based electronic data collection (EDC) system.

PROs will be collected by self-completed questionnaires given to each patient via web-based data collection or telephone interviews. The site will follow up with the patient according to usual practice. Information from the patient's visit may include goniometry and the physician's assessment of treatment outcome and healthcare utilization. Patients will be considered enrolled in the study for a maximum of 4 years post-enrollment or until death, withdrawal of consent, loss to follow-up, or study closure.

ELIGIBILITY:
Inclusion Criteria:

* Women or men 18 years of age or older
* Patients with a Dupuytren's contracture of at least a single joint and a desire for correction
* Patients who are able to read and understand English
* Patients who are capable of understanding and cooperating with the requirements of the study
* Patients who are willing and able to respond to the posttreatment assessments via telephone or internet
* Patients must provide written informed consent, indicating that they understand the purpose of and requirements of the study and are willing to participate in the study.

Exclusion Criteria:

* Patients who decide not to pursue correction of the Dupuytren's contracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community based sample
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The primary objective is to collect real-world data regarding patient reported outcomes of the 3 primary treatment modalities in patients with Dupuytren's contracture. | 4 years

SECONDARY OUTCOMES:
Examine safety, effectiveness and association between treatments and selected healthcare utilization and patient report outcomes. | 4 years
  The secondary objectives are as follows:
  * Examine the safety trends of various treatment options in patients with Dupuytren's contracture
  * Examine the effectiveness trends of various treatment options, specifically evaluating long term contracture recurrence
  * Examine the association between various treatment regimens and healthcare resource utilization
  * Examine the association between various treatments and patient-reported outcomes (PROs) such as disease burden, ADLs, hand functionality, work performance, time to return to work, treatment satisfaction, and patient preference

CONTACTS AND LOCATIONS:
Overall Officials: Urdaneta Veronica, MD, Study Director — Endo Pharmaceuticals
Locations (26):
- United States (26):
  - Raven Orthopaedics, Inc., Burbank, California
  - Core Orthopaedic Medical Center, Encinitas, California
  - Torrey Pines Orthopaedic Medical Group, La Jolla, California
  - Brigid Freyne, MD, Inc., Murrieta, California
  - Hand Surgery Associates, Denver, Colorado
  - Physicians for the Hand, Coral Gables, Florida
  - Florida Medical Research Institute, Lady Lake, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - OrthoGeorgia, Macon, Georgia
  - Rockford Orthopedic Associates, LTD, Rockford, Illinois
  - Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - The Hand Center, Wichita, Kansas
  - Bluegrass Orthopaedics and Hand Care Research, Lexington, Kentucky
  - Faith Regional Health Services, Norfolk, Nebraska
  - The Minimally Invasive Hand Institute, Las Vegas, Nevada
  - Central Jersey Hand Surgery, Eatontown, New Jersey
  - Comprehensive Hand Surgery PC, Brooklyn, New York
  - Beth Isreal Medical Center, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Steadman Hawkins Clinic of the Carolinas, Greenville, South Carolina
  - Core Orthopedics, Sioux Falls, South Dakota
  - The Plastic Surgery Group, Chattanooga, Tennessee
  - OrthoMemphis, Memphis, Tennessee
  - Vanderbilt Orthopaedic Institute, Nashville, Tennessee
  - Charlottesville Orthopaedic Center, PLC, Charlottesville, Virginia